CLINICAL TRIAL: NCT03516487
Title: A Phase 1/2a, First-in-human, Oral Single and Multiple Dose-escalation, Randomized, Double-blinded, Placebo-controlled Study of SYNB1618 in Healthy Adult Volunteers and Adult Subjects With Phenylketonuria to Evaluate Safety, Tolerability, Kinetics, and Pharmacodynamics
Brief Title: Safety and Tolerability of SYNB1618 in Healthy Adult Volunteers and Adult Subjects With Phenylketonuria
Acronym: PKU
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Synlogic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYNB1618-CP-001
Record Dates: First submitted 2018-04-11; First posted 2018-05-04 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Phenylketonuria; Healthy
Keywords: PKU
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Intervention Model Description: Dose-escalating, randomized, double-blinded, placebo-controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- SAD HV: SYNB1618 (1 x 10^10 CFU) (Experimental): HV subjects receive a single oral dose of SYNB1618 (1 x 10^10 colony-forming units [CFU]) in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: SYNB1618
- SAD HV: SYNB1618 (5 x 10^10 CFU) (Experimental): HV subjects receive a single oral dose of SYNB1618 (5 x 10^10 CFU) in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: SYNB1618
- SAD HV: SYNB1618 (1 x 10^11 CFU) (Experimental): HV subjects receive a single oral dose of SYNB1618 (1 x 10^11 CFU) in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: SYNB1618
- SAD HV SB: SYNB1618 (1 x 10^11 CFU) (Experimental): HV subjects receive a single oral dose of SYNB1618 (1 x 10^11 CFU) in a chilled buffered solution on Day 1 in the SAD study (Part 1). On Day 1, subjects in this cohort receive a solid breakfast (SB) that contains approximately the same amount of calories and protein as the meal supplement shake given to subjects in the other SAD cohorts.
  Interventions: Drug: SYNB1618
- SAD HV: SYNB1618 (2 x 10^11 CFU) (Experimental): HV subjects receive a single oral dose of SYNB1618 (2 x 10^11 CFU) in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: SYNB1618
- SAD HV: SYNB1618 (5 x 10^11 CFU) (Experimental): HV subjects receive a single oral dose of SYNB1618 (5 x 10^11 CFU) in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: SYNB1618
- SAD HV: Placebo (Placebo Comparator): HV subjects receive a single oral dose of placebo in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: Placebo
- SAD PKU: SYNB1618 (7 x 10^10 CFU) (Experimental): Subjects with PKU receive a single oral dose of SYNB1618 (7 x 10^10 CFU) in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: SYNB1618
- SAD PKU: Placebo (Placebo Comparator): HV subjects receive a single oral dose of placebo in a chilled buffered solution on Day 1 in the SAD study (Part 1).
  Interventions: Drug: Placebo
- MAD HV: SYNB1618 (1 x 10^10 CFU) (Experimental): HV subjects receive oral SYNB1618 (1 x 10^10 CFU) in a chilled buffered solution 3 times per day (TID) for 7 days in the MAD study (Part 2).
  Interventions: Drug: SYNB1618
- MAD HV: SYNB1618 (5 x 10^10 CFU) (Experimental): HV subjects receive oral SYNB1618 (5 x 10^10 CFU) in a chilled buffered solution TID for 7 days in the MAD study (Part 2).
  Interventions: Drug: SYNB1618
- MAD HV: SYNB1618 (7 x 10^10 CFU) (Experimental): HV subjects receive oral SYNB1618 (7 x 10^10 CFU) in a chilled buffered solution TID for 7 days in the MAD study (Part 2).
  Interventions: Drug: SYNB1618
- MAD HV: SYNB1618 (1 x 10^11 CFU) (Experimental): HV subjects receive oral SYNB1618 (1 x 10^11 CFU) in a chilled buffered solution TID for 7 days in the MAD study (Part 2).
  Interventions: Drug: SYNB1618
- MAD HV: Placebo (Placebo Comparator): HV subjects receive oral placebo in a chilled buffered solution TID for 7 days in the MAD study (Part 2).
  Interventions: Drug: Placebo
- MAD PKU: SYNB1618 (7 x 10^10 CFU) (Experimental): Subjects with PKU receive oral SYNB1618 (7 x 10^10 CFU) in a chilled buffered solution TID for 7 days in the MAD study (Part 2).
  Interventions: Drug: SYNB1618
- MAD PKU: Placebo (Placebo Comparator): Subjects with PKU receive oral placebo in a chilled buffered solution TID for 7 days in the MAD study (Part 2).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SYNB1618 — SYNB1618 is supplied in a buffered solution in 5 mL polypropylene cryovials with a nominal 5 mL fill volume, administered with 100 mL of masking buffer solution.
  Arms: MAD HV: SYNB1618 (1 x 10^10 CFU); MAD HV: SYNB1618 (1 x 10^11 CFU); MAD HV: SYNB1618 (5 x 10^10 CFU); MAD HV: SYNB1618 (7 x 10^10 CFU); MAD PKU: SYNB1618 (7 x 10^10 CFU); SAD HV SB: SYNB1618 (1 x 10^11 CFU); SAD HV: SYNB1618 (1 x 10^10 CFU); SAD HV: SYNB1618 (1 x 10^11 CFU); SAD HV: SYNB1618 (2 x 10^11 CFU); SAD HV: SYNB1618 (5 x 10^10 CFU); SAD HV: SYNB1618 (5 x 10^11 CFU); SAD PKU: SYNB1618 (7 x 10^10 CFU)
Drug: Placebo — Subjects receive placebo orally in a chilled buffered solution (100 mL).
  Arms: MAD HV: Placebo; MAD PKU: Placebo; SAD HV: Placebo; SAD PKU: Placebo

SUMMARY:
This Phase 1/2a, first-in-human, oral single and multiple dose-escalation, randomized, double-blinded, placebo-controlled study is evaluating SYNB1618 in healthy volunteers (HV) and subjects diagnosed with phenylketonuria (PKU), a rare inherited metabolic disorder that occurs in people who are missing an enzyme that the body needs to use phenylalanine (Phe). Eligible subjects receive investigational product (IP) in the clinic and undergo safety monitoring, evaluations, and subsequent follow-up after IP administration.

DETAILED DESCRIPTION:
This study is evaluating the safety, tolerability, kinetics, and pharmacodynamics of SYNB1618 within the following 2 study parts:

Part 1 comprises a single-ascending dose (SAD) study conducted over 4 days in HV male and female subjects in up to 6 dose cohorts (3 treated:1 placebo) to identify the maximum tolerated dose (MTD) within the single-dose range studied. Up to 24 HV subjects are planned for enrollment in this part of the study. Following attainment of the MTD in HV, a SAD cohort of up to 4 subjects (male and female, ≥ 18 years old) previously diagnosed with PKU will be enrolled (3 treated:1 placebo).

Part 2 comprises a multiple-ascending dose (MAD) study conducted in an inpatient setting (6 treated:2 placebo) over 10 days in HV male and female subjects in up to 4 cohorts at doses not exceeding the MTD from the SAD part of the study to identify the MTD of SYNB1618 within the multiple-dose range studied. Up to 32 HV subjects are planned for enrollment in this part of the study. Once the highest MAD cohort and the SAD PKU cohort are completed, a multiple-dose cohort of male and female subjects (≥ 18 years old) previously diagnosed with PKU are evaluated. Up to 20 subjects with PKU are planned for enrollment in the MAD PKU cohort (12 treated:8 placebo).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 to ≤ 64 years.
2. Able and willing to voluntarily complete the informed consent process (subject or subject's representative).
3. Available for and agrees to all study procedures, including feces, urine, and blood collection and adherence to diet control, inpatient monitoring, follow-up visits, and IP ingestion compliance.
4. Male subjects who are sexually abstinent or surgically sterilized (vasectomy), or those who are sexually active with a female partner(s) and agree to use an acceptable method of contraception (such as condom with spermicide) combined with an acceptable method of contraception for their non-pregnant female partner(s) (as defined in Inclusion Criterion #5) after informed consent, throughout the study, and for a minimum of 90 days after the last dose of IP, and who do not intend to donate sperm in the period from screening until 3 months following administration of the investigational medical product.
5. Female subjects that meet one of the following:

   1. Women of childbearing potential must have a negative serum pregnancy test (human chorionic gonadotropin [HCG]) at screening and at baseline prior to the start of IP and must agree to use acceptable method(s) of contraception, combined with an acceptable method of contraception for their male partner(s) (as defined in Inclusion Criterion #4) after informed consent, throughout the study and for a minimum of 90 days after the last dose of IP. Acceptable methods of contraception include hormonal contraception, hormonal or non-hormonal intrauterine device, bilateral tubal occlusion, complete abstinence, vasectomized partner with documented azoospermia 90 days after procedure, diaphragm with spermicide, cervical cap with spermicide, vaginal sponge with spermicide, or male or female condom with or without spermicide.
   2. Premenopausal woman with one of the following: i. Documented hysterectomy; ii. Documented bilateral salpingectomy; iii. Documented bilateral oophorectomy; iv. Documented tubal ligation/occlusion; v. Sexual abstinence is preferred or usual lifestyle of the subject.
   3. Postmenopausal woman (12 months or more amenorrhea verified by follicle stimulating hormone assessment and over 45 years of age in the absence of other biological or physiological causes).
6. Screening laboratory evaluations (e.g., chemistry panel, complete blood count with differential, prothrombin time/activated partial thromboplastin time, urinalysis, C reactive protein, creatinine clearance) and electrocardiogram must be within normal limits or judged to be not clinically significant by the Investigator.
7. Stable diet including protein intake for at least 60 days prior to screening assessments.
8. Able to produce at least 2 bowel movements per week on average without the assistance of laxatives.

   In addition to the above criteria for HV, inclusion criteria for PKU subjects are as noted below.
9. Diagnosis of classic PKU by either medical history of blood Phe concentration of >1200 µmol/L at any time OR genetic diagnosis.
10. Blood Phe concentration of ≥ 600 µmol/L at Screening.
11. Stable diet including stable medical formula regimen (if used) for 60 days prior to screening assessments.

Exclusion Criteria:

1. Acute or chronic medical, surgical, psychiatric, or social condition or laboratory abnormality that may increase subject risk associated with study participation, compromise adherence to study procedures and requirements, or confound interpretation of study safety or pharmacodynamic results and, in the judgment of the Investigator, make the subject inappropriate for enrollment.
2. Body mass index < 18.5 or ≥ 30 kg/m^2 (> 40 kg/m^2 for PKU subjects).
3. History of or current immunodeficiency disorder including autoimmune disorders and human immunodeficiency virus antibody positivity.
4. Hepatitis B surface antigen positivity (subjects with hepatitis B surface antibody positivity and hepatitis B core antibody positivity are not excluded, provided that the hepatitis B surface antigen is negative).
5. Hepatitis C antibody positivity, unless a hepatitis C virus ribonucleic acid test is performed and the result is negative.
6. History of febrile illness, confirmed bacteremia, or other active infection within 30 days prior to the anticipated first dose of IP.
7. History of active or chronic passage of 3 or more loose stools per day.
8. Active laxative use within 30 days prior to the anticipated first dose of IP.
9. Active inflammatory or irritable bowel disorder of any grade.
10. Active or past history of gastrointestinal bleeding within 60 days prior to the Screening Visit as confirmed via hospitalization-related event(s) or medical history of hematemesis or hematochezia.
11. Intolerance of or allergic reaction to E. coli Nissle or any of the ingredients in SYNB1618 or placebo formulations.
12. Any condition, prescription medication, or over-the-counter product that may possibly affect absorption of medications or nutrients (e.g., celiac disease, gastrectomy, bypass surgery, ileostomy).
13. Currently taking or plans to take any type of systemic (e.g., oral or intravenous) antibiotic within 28 days prior to the anticipated first dose of IP through the final outpatient follow-up. Exception: topical antibiotics are allowed.
14. Major surgery (an operation upon an organ within the cranium, chest, abdomen, or pelvic cavity) or inpatient hospital stay within the 3 months prior to the anticipated first dose of IP.
15. Planned surgery, hospitalizations, dental, or interventional studies between screening and last anticipated visit that might require antibiotics.
16. Taking or planning to take probiotic supplements (enriched foods excluded) within 28 days prior to the anticipated first dose of IP and for the duration of participation and follow-up.
17. Dependence on drugs of abuse.
18. Regular alcohol consumption in excess of 14 standard drinks/week for men and in excess of 7 standard drinks/week for women and/or any evidence of binge or heavy drinking (according to National Institute on Alcohol Abuse and Alcoholism guidelines). One drink is equivalent to 12 g of alcohol: 12 oz (360 mL) of beer, 5 oz (150 mL) of wine or 1.5 oz (45 mL) of 80 proof distilled spirits.
19. Administration or ingestion of an investigational drug within 60 days or 5 half-lives, whichever is longer, prior to the Screening Visit or current enrollment in an investigational study. (PKU subjects who participate in the PKU SAD cohort may be eligible for screening for the PKU MAD cohort ≥ 30 days after the last dose of IP.)
20. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular (including stable coronary artery disease/angina or prior cardiac stent), hepatic, neurologic, or allergic disease including drug allergies.
21. Screening laboratory parameters within the acceptable range.

    In addition to the above criteria for HV, exclusion criteria for PKU subjects are as noted below.
22. Currently taking (within 1 week prior to screening) sapropterin (KUVAN®).
23. Currently taking (within 6 months prior to screening) pegylated recombinant phenylalanine ammonia lyase (PALYNZIQ™).
24. History of a severe immune reaction based on National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) after administration of pegylated recombinant phenylalanine ammonia lyase (PALYNZIQ).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-04-17 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Number of Subjects With Treatment-Emergent Adverse Events | Up to 4 months
  Toxicity is graded in accordance with the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 4.03. Adverse events (AEs) are reported based on clinical laboratory tests, vital sign and weight measurements, physical examinations, electrocardiograms, and any other medically indicated assessments, including subject interviews, from the time informed consent is signed through the end of the safety follow-up period.
  AEs are considered to be treatment emergent (TEAE) if they occur or worsen in severity after the first dose of study treatment. TEAEs are considered treatment-related if relationship to study drug is possibly related, probably related, or definitely related.

SECONDARY OUTCOMES:
Clearance of SYNB1618 From Feces | Up to 4 months
  SYNB1618 transit through the gastrointestinal tract is measured with fecal quantitative polymerase chain reaction (qPCR) assays from fecal samples collected at baseline, daily during the dosing period, at the time of discharge from the inpatient unit, and weekly thereafter for up to 8 weeks after the last dose of investigational product (IP) until a subject has a negative SYNB1618 fecal test. SYNB1618 clearance reflects a test value of below the limit of quantitation (BLQ) occurring after the indicated number of days following the last dose of IP.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - PRA Health Sciences, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Puurunen MK, Vockley J, Searle SL, Sacharow SJ, Phillips JA 3rd, Denney WS, Goodlett BD, Wagner DA, Blankstein L, Castillo MJ, Charbonneau MR, Isabella VM, Sethuraman VV, Riese RJ, Kurtz CB, Brennan AM. Safety and pharmacodynamics of an engineered E. coli Nissle for the treatment of phenylketonuria: a first-in-human phase 1/2a study. Nat Metab. 2021 Aug;3(8):1125-1132. doi: 10.1038/s42255-021-00430-7. Epub 2021 Jul 22. PMID 34294923
- [Derived] Charbonneau MR, Denney WS, Horvath NG, Cantarella P, Castillo MJ, Puurunen MK, Brennan AM. Development of a mechanistic model to predict synthetic biotic activity in healthy volunteers and patients with phenylketonuria. Commun Biol. 2021 Jul 22;4(1):898. doi: 10.1038/s42003-021-02183-1. PMID 34294862